CLINICAL TRIAL: NCT06995820
Title: A Phase I Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of AZD1613 Following Single and Multiple Dose Administration in Healthy Participants
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of AZD1613 in Healthy Participants.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D9050C00001
Record Dates: First submitted 2025-05-28; First posted 2025-05-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Single ascending dose; Multiple ascending dose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A1 (SAD): AZD1613 (Dose 1) SC (Experimental): Participants will receive a single dose of AZD1613 (Dose 1) or matching placebo to AZD1613 as SC injection on Day 1.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part A1 (SAD): AZD1613 (Dose 2) SC (Experimental): Participants will receive a single dose of AZD1613 (Dose 2) or matching placebo to AZD1613 as SC injection on Day 1.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part A1 (SAD): AZD1613 (Dose 3) SC (Experimental): Participants will receive a single dose of AZD1613 (Dose 3) or matching placebo to AZD1613 as SC injection on Day 1.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part A1 (SAD): AZD1613 (Dose 4) SC (Experimental): Participants will receive a single dose of AZD1613 (Dose 4) or matching placebo to AZD1613 as SC injection on Day 1.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part A1 (SAD): AZD1613 (Dose 5) IV (Experimental): Participants will receive a single dose of AZD1613 (Dose 5) or matching placebo to AZD1613 as an IV infusion on Day 1.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part A1 (SAD): AZD1613 (Dose 6) IV (Experimental): Participants will receive a single dose of AZD1613 (Dose 6) or matching placebo to AZD1613 as an IV infusion on Day 1.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part A2 (SAD): AZD1613 (Dose 7) SC or IV (Chinese) (Experimental): Chinese participants will receive a single dose of AZD1613 (Dose 7) or matching placebo to AZD1613 as SC injection or IV infusion on Day 1.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part A3 (SAD): AZD1613 (Dose 8) SC or IV (Japanese) (Experimental): Japanese participants will receive a single dose of AZD1613 (Dose 8) or matching placebo to AZD1613 as SC injection or IV infusion on Day 1.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part A3 (SAD): AZD1613 (Dose 9) SC or IV (Japanese) (Experimental): Japanese participants will receive a single dose of AZD1613 (Dose 9) or matching placebo to AZD1613 as SC injection or IV infusion on Day 1.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part B (MAD): AZD1613 (Dose 10) SC (Experimental): Participants will receive multiple doses of AZD1613 (Dose 10) or matching placebo to AZD1613 as SC injection or IV infusion on Days 1, 29 and 57.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part B (MAD): AZD1613 (Dose 11) SC (Experimental): Participants will receive multiple doses of AZD1613 (Dose 11) or matching placebo to AZD1613 as SC injection or IV infusion on Days 1, 29 and 57.
  Interventions: Drug: AZD1613; Drug: Placebo
- Part B (MAD): AZD1613 (Dose 12) IV (Experimental): Participants will receive multiple doses of AZD1613 (Dose 12) or matching placebo to AZD1613 as an IV infusion on Days 1, 29 and 57.
  Interventions: Drug: AZD1613; Drug: Placebo

INTERVENTIONS:
Drug: AZD1613 — AZD1613 will be administered as either SC injection or IV infusion on Day 1 in Part A and on Days 1, 29 and 57 in Part B of the study.
Drug: Placebo — Placebo will be administered as either SC injection or IV infusion on Day 1 in Part A and Days 1, 29 and 57 in Part B fo the study.

SUMMARY:
The purpose of the study is to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of AZD1613 in healthy participants, including Japanese and Chinese descent.

DETAILED DESCRIPTION:
This is a first-in-human, randomized, single-blind, placebo-controlled, single and multiple ascending dose study in healthy participants and will be conducted at a single study center. It consists of two parts: Part A (Single Ascending Dose - SAD) and Part B (Multiple Ascending Dose - MAD).

Part A of the study is a SAD sequential group design study and will consist of Parts A1, A2, and A3. Part A1 is planned to consist of 6 cohorts, Part A2 is planned to consist of one cohort of participants of Chinese descent, and Part A3 is planned to consist of 2 cohorts of participants of Japanese descent.

Parts A1, A2, and A3 of the study will comprise of:

1. A Screening Period of maximum 28 days.
2. A Treatment Period during which each participant will receive a single subcutaneous (SC) or intravenous (IV) dose of either AZD1613 or placebo on Day 1.
3. A Follow-up Period where participants will return to the study center for non-residential visits until Day 105.

Part B of the study will be a MAD sequential group design study. Up to 3 dose levels of AZD1613 are planned to be investigated in 3 cohorts of healthy participants.

Part B of the study will comprise of:

1. A Screening Period of maximum 28 days.
2. Three Treatment Periods during which participants will receive 3 single subcutaneous (SC) or intravenous (IV) doses of AZD1613 or placebo at 28-day intervals (Day 1, Day 29, and Day 57).
3. A Follow-up Period where participants will return to the study center for non-residential visits until Day 161.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females of non-childbearing potential with suitable veins for cannulation or repeated venipuncture.
2. Negative pregnancy test at screening and admission (females only).
3. Females of non-childbearing potential confirmed by postmenopausal status or irreversible surgical sterilization.
4. Sexually active fertile males must use contraception methods from first administration until 3 months after the last follow-up visit.
5. Body mass index (BMI) between 18 and 32 kg/m² and weight at least 50 kg.
6. Participants of Chinese descent (Part A2) must have both parents and four grandparents who are Chinese.
7. Participants of Japanese descent (Part A3) must have both parents and four grandparents who are Japanese.

Exclusion Criteria:

1. The history of any clinically important disease or disorder may either put the participant at risk due to participation in the study, influence the results, or affect the participant's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic, or renal disease affecting drug absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of first administration.
4. Abnormal lab values at screening or admission (e.g., alanine aminotransferase (ALT) > upper limit normal (ULN), aspartate aminotransferase (AST) > ULN, bilirubin > 1.5 × ULN, estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73 m², hemoglobin < lower limit normal [LLN]).
5. Any clinically important abnormalities in clinical chemistry, hematology, or urinalysis results.
6. Any positive result for serum Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), Hepatitis C virus antibody (HCV Ab) or Human immunodeficiency virus (HIV).
7. Abnormal vital signs after 5 minutes supine rest at screening or admission (e.g., systolic BP < 90 mmHg or ≥ 140 mmHg, diastolic BP < 50 mmHg or ≥ 90 mmHg, heart rate < 45 or > 85 bpm).
8. Any clinically important abnormalities in rhythm, conduction, or morphology of resting 12-lead Electrocardiogram (ECG) at screening or admission (e.g., prolonged QTcF > 450 ms, shortened QTcF < 340 ms, family history of long QT syndrome).
9. Smokers who smoke more than 5 cigarettes per day and cannot adhere to no smoking during residential visits.
10. Known or suspected history of alcohol or drug abuse or excessive alcohol intake.
11. Positive screen for drugs of abuse or alcohol at screening or admission.
12. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
13. Use of prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, or intake of > 3 × daily recommended levels of vitamins and minerals during the 2 weeks prior to first administration.
14. Plasma donation within one month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening.
15. Received another new chemical entity within 30 days or 5 half-lives (whichever is longest) of first administration.
16. Previously received AZD1613.
17. Involvement in the planning and/or conduct of the study.
18. Judgment by the Investigator that the participant should not participate due to minor medical complaints or non-compliance with study procedures.
19. Medical dietary restrictions or inability/unwillingness to comply with meals provided during the stay at the Clinical Unit.
20. Inability to communicate reliably with the Investigator.
21. Vulnerable participants (e.g., kept in detention, protected adults under guardianship).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2026-09-23 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious AEs. | AEs: Part A: From Day 1 to Final Follow-up (Day 105); Part B: From Day 1 to Final Follow-up (Day 161); SAEs: Part A: From Screening (Day -28 to Day -2) to Final Follow-up visit (Day 105) Part B: From Screening (Day -28) to Final Follow-up visit (Day 161)
  To assess the safety and tolerability of AZD1613 following SC and/or IV administration of single and multiple ascending doses.

SECONDARY OUTCOMES:
Area under concentration-time curve from time 0 to infinity (AUCinf) (Day 1 only) | Part A: From Day 1 (pre-dose) to Day 105; Part B: From Day 1 (pre-dose) to Day 141
  To characterize the single and multiple dose PK of AZD1613 following SC and/or IV administration.
Area under concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | Part A: From Day 1 (pre-dose) to Day 105; Part B: From Day 1 (pre-dose) to Day 141
  To characterize the single and multiple dose PK of AZD1613 following SC and/or IV administration.
Maximum observed drug concentration (Cmax) | Part A: From Day 1 (pre-dose) to Day 105; Part B: From Day 1 (pre-dose) to Day 141
  To characterize the single and multiple dose PK of AZD1613 following SC and/or IV administration.
Incidence of positive anti-drug antibodies (ADAs) against AZD1613 in serum | Part A: Day 1 (pre-dose), Day 29, Day 57 and Day 105; Part B: Day 1 (pre-dose), Day 29 (pre-dose), Day 57 (pre-dose), Day 85 and Day 161
  To evaluate the immunogenecity of AZD1613.
Change from baseline in study-specific biomarker ABC | Part A: From Day 1 to Day 105; Part B: From Day -1 to Day 161
  To evaluate target engagement by assessing change in plasma biomarker.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/